CLINICAL TRIAL: NCT01418573
Title: Glycemic Response After Two Palaeolithic-type Meals Compared to a Modern-type Meal Composed According to WHO Guidelines
Brief Title: Glycemic Response After Palaeolithic-type Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Leatherhead Food Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FDS-BNH-0100
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2012-02

CONDITIONS: Glycemic Index of a Meal
Keywords: glucose, insulin, post prandial
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Palaeolithic-type meal 1 (Experimental)
  Interventions: Other: Palaeolithic meal 1
- Palaeolithic-type meal 2 (Experimental)
  Interventions: Other: Palaeolithic meal 2
- The reference meal (Placebo Comparator)
  Interventions: Other: Reference meal

INTERVENTIONS:
Other: Palaeolithic meal 1 — Based on estimated ratios for protein, fat and carbohydrates that are typical of Hunter-Gatherers and does not contain ingredients that were not available in pre-neolithic times
  Arms: Palaeolithic-type meal 1
Other: Palaeolithic meal 2 — Based on WHO dietary guidelines for protein, fat and carbohydrate but does not contain ingredients that were not available in pre neolithic times
  Arms: Palaeolithic-type meal 2
Other: Reference meal — Based on WHO dietary guidelines for protein, fat and carbohydrate.
  Arms: The reference meal

SUMMARY:
The objective of the study is to show post-prandial benefits of Palaeolithic-type meals as compared to a meal constructed along the lines of the WHO dietary recommendations.

DETAILED DESCRIPTION:
The effects of this set of meals will be assessed with respect to blood

* blood glucose
* plasma insulin
* satiety scores
* plasma gut hormones It is hypothesised that lower post prandial blood glucose concentration, a lower insulin response and increased satiety will be seen after the Palaeolithic meals compared with a reference meal

ELIGIBILITY:
Inclusion Criteria:

* male
* ≥ 18 and ≤ 60 years old
* Body mass index (BMI) ≥ 18 and ≤ 27.0 kg/m2
* Apparently healthy
* Not smoking
* A fasting blood glucose value within the normal reference value

Exclusion Criteria:

- No prescribed medication

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 0-2 hours
  positive incremental area under the concentration versus time
Plasma insulin | 0-2 hours
  net incremental area under the curve
Peak blood glucose | 0-2 hours
  maximal blood glucose value

SECONDARY OUTCOMES:
Satiety scores | 0-2 hours
  area under the curve
Gut hormone panel | 0-3 hours
  Average concentration over time

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Pombo, Principal Investigator — Leatherhead Food Research
Locations (1):
- Leatherhead Food Research, Leatherhead, Surrey, United Kingdom

REFERENCES:
- [Background] Frassetto LA, Schloetter M, Mietus-Synder M, Morris RC Jr, Sebastian A. Metabolic and physiologic improvements from consuming a paleolithic, hunter-gatherer type diet. Eur J Clin Nutr. 2009 Aug;63(8):947-55. doi: 10.1038/ejcn.2009.4. Epub 2009 Feb 11. PMID 19209185
- [Background] Jonsson T, Granfeldt Y, Ahren B, Branell UC, Palsson G, Hansson A, Soderstrom M, Lindeberg S. Beneficial effects of a Paleolithic diet on cardiovascular risk factors in type 2 diabetes: a randomized cross-over pilot study. Cardiovasc Diabetol. 2009 Jul 16;8:35. doi: 10.1186/1475-2840-8-35. PMID 19604407
- [Derived] Bligh HF, Godsland IF, Frost G, Hunter KJ, Murray P, MacAulay K, Hyliands D, Talbot DC, Casey J, Mulder TP, Berry MJ. Plant-rich mixed meals based on Palaeolithic diet principles have a dramatic impact on incretin, peptide YY and satiety response, but show little effect on glucose and insulin homeostasis: an acute-effects randomised study. Br J Nutr. 2015 Feb 28;113(4):574-84. doi: 10.1017/S0007114514004012. Epub 2015 Feb 9. PMID 25661189